CLINICAL TRIAL: NCT04575896
Title: An Open-label, Non-randomized Pilot Study to Determine the Safety and Efficacy of Two Weeks of Fixed-dose Glecaprevir and Pibrentasvir as Pre- and Post-exposure Prophylactic Therapy
Brief Title: Kidney Transplants in Hepatitis C Negative Recipients With Hepatitis C Viremic Donors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00237097
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: End Stage Renal Disease; Hepatitis C
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Deceased donor HCV RNA PCR+ (Experimental): Participants who receive a kidney from HCV RNA PCR + deceased donor will receive glecaprevir/pibrentasvir 300 mg/120 mg once daily by mouth for 2 weeks
  Interventions: Drug: Glecaprevir/pibrentasvir

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — Glecaprevir/pibrentasvir 300mg/120mg once daily by mouth for 2 weeks post-transplant.
  Other Names: Mavyret

SUMMARY:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Treatment will include glecaprevir 300 mg / pibrentasvir 120 mg (G-P) administered on-call to the operating room for the renal transplant procedure and continued for 2 weeks post-renal transplant.

DETAILED DESCRIPTION:
In this study, individuals without hepatitis C infection who are on the kidney transplant waitlist will receive a kidney from a deceased donor with hepatitis C infection and will be treated for hepatitis C at the same time. Treatment will include glecaprevir 300 mg / pibrentasvir 120 mg (G-P) administered on-call to the operating room for the renal transplant procedure and continued for 2 weeks post-renal transplant. The participant will continue to be tested for Hepatitis C for 12 weeks post-treatment.

The primary hypothesis is that prophylactic treatment with glecaprevir/pibrentasvir before and after transplant will prevent the establishment of HCV infection in the recipients of kidneys from HCV-infected deceased donors. Based on the success of preliminary studies, the objective of the study is to evaluate the safety and efficacy of 2 weeks of G-P as prophylaxis for HCV D+/R- kidney transplant.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Participants ≥ 18 years old
* On the deceased donor kidney waitlist at Johns Hopkins Hospital
* Awaiting a first or second kidney transplant
* No available living kidney donors
* On hemodialysis or peritoneal dialysis or stage 5 chronic kidney disease (CKD) defined as a glomerular filtration rate <15 ml/min for ≥ past 90 days
* HCV-uninfected (by both antibody and RNA PCR) and without any behavioral risk factors for contracting HCV other than being on hemodialysis
* Calculated panel reactive anti-human leukocyte antigens (anti-HLA) antibody (flow cPRA) below 80%

Recipient Exclusion Criteria:

* Plan to receive a multi-organ transplant
* Plan to receive a dual kidney transplant (including en bloc)
* History of prior solid organ transplant other than first kidney transplant
* Participating in another study that involves an intervention or investigational product
* Plan to receive a blood type incompatible kidney
* History of human immunodeficiency (HIV), hepatitis C (HCV), or active hepatitis B (HBV) infection, defined as being on active antiviral treatment for HBV, detectable hepatitis B surface Ag or detectable hepatitis B DNA
* Unable to safely substitute or discontinue a medication that is contraindicated with the study medication
* Psychiatric or physical illness that in the opinion of the investigator would make it unsafe to proceed with transplantation or interfere with the ability of the subject to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Desai, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Durand CM, Barnaba B, Yu S, Brown DM, Chattergoon MA, Bair N, Naqvi FF, Sulkowski M, Segev DL, Desai NM. Four-Week Direct-Acting Antiviral Prophylaxis for Kidney Transplantation From Hepatitis C-Viremic Donors to Hepatitis C-Negative Recipients: An Open-Label Nonrandomized Study. Ann Intern Med. 2021 Jan;174(1):137-138. doi: 10.7326/M20-1468. Epub 2020 Sep 8. No abstract available. PMID 32894697

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deceased Donor HCV RNA PCR+
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2
  Race: Black | 5
  Race: White | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Viral Response as Assessed by Number of Participants With Undetectable Hepatitis C RNA
Description: This is the number of participants with undetectable hepatitis C RNA in the blood at 12 weeks after stopping treatment (Number of kidney transplant recipients with HCV RNA < Lower Limit Of Quantification (LLOQ)).
Time Frame: 12 weeks after completing therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Deceased Donor HCV RNA PCR+
Number analyzed (Participants) | 10
Participants | 10

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Deceased Donor HCV RNA PCR+
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deceased Donor HCV RNA PCR+ (N=10)
urinary tract infection (Renal and urinary disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
right iliac hematoma (Renal and urinary disorders) | 1 (1)
hypotension (orthostatic) (General disorders) | 1 (1)
creatinine increased (Renal and urinary disorders) | 1 (1)
hyperkalemia (Renal and urinary disorders) | 2 (2)
acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deceased Donor HCV RNA PCR+ (N=10)
fever (General disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
hyperkalemia (Renal and urinary disorders) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
dialysis access malfunction (Renal and urinary disorders) | 1 (1)
flash pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Our study is limited by the small sample size and single-group design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/96/NCT04575896/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT04575896/ICF_001.pdf